CLINICAL TRIAL: NCT03097328
Title: A Phase II Study of TAK-228 In Patients With Previously Treated Metastatic Renal Cell Carcinoma
Brief Title: Study of TAK-228 In Patients With Previously Treated Metastatic Renal Cell Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bradley A. McGregor, MD (Other)
Collaborators: Calithera Biosciences, Inc (Industry)
Responsible Party: Sponsor-Investigator, Bradley A. McGregor, MD, Sponsor Investigator, Dana-Farber Cancer Institute
Organization: Dana-Farber Cancer Institute (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16-527
Record Dates: First submitted 2017-03-15; First posted 2017-03-31 (Actual); Results first posted 2022-02-24 (Actual); Last update posted 2024-04-29 (Actual); Status verified 2024-04

CONDITIONS: Renal Cell Carcinoma
Keywords: Renal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — sapanisertib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- TAK-228 (Experimental): * TAK-228 will be taken orally on a weekly basis for 4 weeks per cycle
  * Dosage will be determined by the study team
  Interventions: Drug: TAK-228

INTERVENTIONS:
Drug: TAK-228 — TAK-228 works to inhibit or interfere with cellular functions involved in cell growth and survival. TAK-228 specifically targets a type of protein that can make chemicals that trigger cell growth, including cancer cell growth
  Other Names: INK128

SUMMARY:
This research study is investigating a drug as a possible treatment for metastatic renal cell carcinoma. The intervention involved in this study is TAK-228.

DETAILED DESCRIPTION:
This research study is a Phase II clinical trial. Phase II clinical trials test the safety and effectiveness of an investigational intervention to learn whether the intervention works in treating a specific disease. "Investigational" means that the intervention is being studied.

The FDA (the U.S. Food and Drug Administration) has not approved TAK-228 as a treatment for any disease but it is being investigated as a treatment for advanced solid tumors, blood disorders, and inflammatory diseases. TAK-228 works to inhibit or interfere with cellular functions involved in cell growth and survival. TAK-228 specifically targets a type of protein that can make chemicals that trigger cell growth, including cancer cell growth. This protein may also cause cells to produce proteins that trigger the development of new blood vessels. Cancers need new blood vessels in order to grow. In some types of cancer, this type of protein (mTOR) is switched on, and it makes the cancer cells grow and produce new blood vessels. mTOR blockers (inhibitors) are a newer type of cancer growth blocker that can stop the growth of some types of cancer.

Researchers hope to learn how participants with previously treated mRCC will respond to treatment with TAK-228. Other goals of this study include assessing the types of side effects associated TAK-228 and whether there is a relationship between certain genetic mutations (changes to your DNA) and participant responses to the drug.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Measurable disease according to RECIST 1.1 within 28 days prior to registration.
* Documented pathologic diagnosis of RCC. All subtypes eligible including but not limited to clear cell, papillary, chromophobe, collecting duct carcinoma, medullary carcinoma, and unclassified categories. Sarcomatoid and rhabdoid differentiation are allowed.
* Patients with clear cell histology must have demonstrated: 1) Progression on at least one prior anti -angiogenic agent unless intolerable; AND 2) progression on at least one agent that blocks the PD-1 pathway unless felt by the treating physician to be contraindicated (examples include but are not limited to: patients with autoimmune disease or patients requiring systemic steroids greater than 10 mg/day prednisone or its equivalent) or if they have been discontinued due to toxicity. Prior rapalogues are allowed.
* Patients with non-clear cell histology must have received at least one prior anti-cancer therapy. Prior rapalogues are allowed.
* Left ventricular ejection fraction (LVEF) ³ lower limit of normal (LLN) as assessed by either multigated acquisition (MUGA) scan or echocardiogram (ECHO).
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2.
* Must have adequate organ and bone marrow function.
* Hematological

  * Absolute Neutrophil Count (ANC) ≥ 1500 K/mm^3 (without use of G-CSF 4 weeks prior to enrollment)
  * Hemoglobin (Hgb) ≥ 9 g/dL (transfusions allowed)
  * Platelets (Plts) ≥ 100 k/mm^3
* Renal

  * Calculated creatinine clearance (Cockcroft-Gault formula will be used to calculate creatinine clearance) ≥ 30 mL/min
  * Urinalysis: For patients with 2+ proteinuria on urinalysis, 24 hour urine collection should be obtained, 24 hour urine protein should be <2 grams.
* Hepatic

  * Bilirubin ≤ 1.5 × upper limit of normal (ULN). For subjects with Gilbert's disease ≤ 3.0 mg/dL
  * Aspartate aminotransferase (AST) ≤ 2.5 × ULN; ≤ 5 x ULN if liver metastases are present
  * Alanine aminotransferase (ALT) ≤ 2.5 × ULN; ≤ 5 x ULN if liver metastases are present
* Metabolic

  * Glycosylated hemoglobin (HbA1c) < 7.0%,
  * Fasting serum glucose ≤ 130 mg/dL
  * Fasting triglycerides ≤ 300 mg/dL
* Recovery to baseline or ≤ grade 1 Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 from toxicities related to any prior treatment, unless adverse events are clinically non-significant and/or stable on supportive therapy.
* Capable of understanding and complying with the protocol requirements and has signed the informed consent document. Voluntary written consent must be given before performance of any study related procedure not part of standard medical care, with the understanding that consent may be withdrawn by the subject at any time without prejudice to future medical care.
* Submission of formalin-fixed, paraffin-embedded (FFPE) archival tumor specimens from the previous 18 months, if available. If not available, a fresh tumor biopsy prior to treatment initiation is MANDATORY unless determined medically unsafe or not feasible by the site investigator.

  * The archival specimen must contain adequate viable tumor tissue.
  * Specimens may consist of a tissue block (preferred and should contain the highest grade of tumor) or a recommended minimum of 20 unstained serial sections. Fine-needle aspiration, brushings, cell pellet from pleural effusion, bone marrow aspirate/biopsy are not acceptable.
  * Distant metastases specimens are preferred but if not available primary nephrectomy specimens are acceptable.
* Subjects who experience a disease response per RECIST 1.1 criteria followed by subsequent progression will be required to have a post-treatment biopsy if feasible and safe.
* Sexually active subjects and their partners must agree to use medically accepted methods of contraception.

  * For women:

    * Postmenopausal for at least 1 year before the screening visit, OR
    * Surgically sterile, OR
    * Agree to practice 1 effective method of contraception and 1 additional effective (barrier) method at the same time, from the time of signing the informed consent through 90 days (or longer, as mandated by local labeling [eg. USPI, SmPC, etc.] after the last dose of study drug, OR
    * Agree to practice true abstinence, when this is in line with the preferred and usual lifestyle of the subject (Periodic abstinence [e.g, calendar, ovulation, symptothermal, postovulation methods] and withdrawal, spermicides only, and lactational amenorrhea are not acceptable methods of contraception. Female and male condoms should not be used together.)
  * For men:

    * Even if surgically sterilized (ie, status post-vasectomy), they must agree to practice highly effective barrier contraception during the entire study treatment period and through 120 days after the last dose of study drug, OR
    * Agree to practice true abstinence, when this is in line with the preferred and usual lifestyle of the subject (Periodic abstinence [e.g, calendar, ovulation, symptothermal, postovulation methods for the female partner] and withdrawal, spermicides only, and lactational amenorrhea are not acceptable methods of contraception. Female and male condoms should not be used together.)
    * Agree not to donate sperm during the course of this study or 120 days after receiving their last dose of study drug

Exclusion Criteria:

* Subjects with a history of deep vein thrombosis (DVT) or pulmonary embolism (PE) within 6 months of study treatment initiation.
* Receipt of any type of small molecular kinase inhibitor (including investigational kinase inhibitors) within 2 weeks of enrollment or receipt of any anti-cancer therapy (including investigational therapy, monoclonal antibodies, cytokine therapy) within 3 weeks of enrollment.
* Treatment with any investigational products within 3 weeks before the first dose of study drug.
* Radiation therapy for bone metastases within 2 weeks, other external radiation therapy within 4 weeks of enrollment.
* Received prior hemibody external radiotherapy.
* Known brain metastases or cranial epidural disease unless adequately treated with radiotherapy, radiosurgery, or surgery and stable for at least 4 weeks prior to enrollment as documented by magnetic resonance imaging (MRI) or computed tomography (CT) imaging. Treated brain metastases are defined as having no ongoing requirement for steroids and no evidence of progression or hemorrhage after treatment for at least 4 weeks prior to enrollment as documented by MRI or CT imaging.
* Imminent or established spinal cord compression based on clinical and/or imaging. In subjects with untreated imminent or established spinal cord compression, treatment with standard of care as clinically indicated should be completed at least 4 weeks before enrollment.
* The subject has a history of any of the following within the last 6 months before administration of the first dose of the drug:

  * Ischemic myocardial event, including angina requiring therapy and artery revascularization procedures
  * Ischemic cerebrovascular event, including transient ischemic attack and artery revascularization procedures
  * Requirement for inotropic support (excluding digoxin) or serious (uncontrolled) cardiac arrhythmia (including atrial flutter/fibrillation, ventricular fibrillation or ventricular tachycardia)
  * Placement of a pacemaker for control of rhythm
  * New York Heart Association (NYHA) Class III or IV heart failure
  * Significant active cardiovascular or pulmonary disease including:

    * Uncontrolled hypertension defined as sustained BP >160 mm Hg systolic or > 95 mm Hg diastolic despite optimal antihypertensive treatment.
    * Pulmonary hypertension
    * Uncontrolled asthma or O2 saturation < 90% by arterial blood gas analysis or pulse oximetry on room air
    * Significant valvular disease; severe regurgitation or stenosis by imaging independent of symptom control with medical intervention, or history of valve replacement
    * History of arrhythmia requiring an implantable cardiac defibrillator
    * Medically significant (symptomatic) bradycardia
* Poorly controlled diabetes mellitus defined as glycosylated hemoglobin (HbA1c) > 7%; subjects with a history of transient glucose intolerance due to corticosteroid administration may be enrolled in this study if all other inclusion/exclusion criteria are met
* Active gastrointestinal (GI) disorders including those associated with a high risk of perforation or fistula formation. Subjects with enteric stomata (such as ileostomy, colostomy) are also excluded:
* Tumors invading the GI-tract, active peptic ulcer disease, inflammatory bowel disease, diverticulitis, cholecystitis, symptomatic cholangitis or appendicitis, acute pancreatitis or acute obstruction of the pancreatic or biliary duct, or gastric outlet obstruction.

  --Abdominal fistula, gastrointestinal perforation, bowel obstruction, or intraabdominal abscess within 12 weeks before enrollment. NOTE: Complete healing of an intra-abdominal abscess must be confirmed before enrollment.
* Clinically significant hematemesis or hemoptysis of > 0.5 teaspoon (2.5 ml) of red blood, or other history of significant bleeding (such as pulmonary hemorrhage) within 4 weeks of enrollment.
* Other clinically significant disorders such as:

  * Known active infection requiring systemic treatment, infection with human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS)-related illness, chronic hepatitis B or known or suspected active hepatitis C infection.
  * Serious non-healing wound or ulcer.
  * Malabsorption syndrome.
  * Symptomatic hypothyroidism.
  * Moderate to severe hepatic impairment (Child-Pugh B or C).
  * Requirement for hemodialysis or peritoneal dialysis.
  * History of solid organ transplantation.
* Major surgery (such as GI surgery) within 6 weeks of enrollment. However, subjects who have had a nephrectomy may be enrolled 4 weeks after surgery, providing there are no wound-healing complications. Subjects with clinically relevant ongoing complications from prior surgery are not eligible. The following are not considered to be major procedures: Thoracentesis, paracentesis, port placement, laparoscopy, thoracoscopy, bronchoscopy, endoscopic ultrasonographic procedures, mediastinoscopy, skin biopsies, incisional biopsies, imaging-guided biopsy for diagnostic purposes, and routine dental procedures.
* QTcF (Fridericia formula for the QT interval correction for the heart rate) > 480 msec within 4 weeks of enrollment. If the initial QTcF is found to be > 480 msec, two additional electrocardiograms (EKGs) separated by at least 3 minutes should be performed. If the average of these three consecutive results for QTcF is ≤ 480 msec, the subject meets eligibility in this regard. Subjects with history of congenital long QT syndrome, or torsades de pointes, are not allowed.
* Pregnant or lactating females.
* Inability to swallow tablets or capsules.
* Previously identified allergy or hypersensitivity to components of the study treatment formulations.
* Malignancies other than RCC within 5 years of first study treatment with the exception of those with negligible risk of metastases or death (carcinoma in situ of the cervix, basal or squamous cell skin cancer, localized prostate cancer, ductal carcinoma in situ of the breast, non-muscle invasive urothelial carcinoma).
* Any serious medical or psychiatric illness that could, in the site investigator's opinion, potentially interfere with the completion of treatment according to this protocol.
* Daily or chronic use of a proton pump inhibitor (PPI) and/or having taken a PPI within 7 days before receiving the first dose of study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2021-07-20 (Actual); Study Completion 2024-04-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bradley McGregor, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (8):
- United States (8):
  - University of California, San Diego Moores Cancer Center, La Jolla, California
  - University of Colorado Cancer Center, Aurora, Colorado
  - University of Chicago Medical Center, Chicago, Illinois
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - University of Minnesota, Minneapolis, Minnesota

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] McGregor BA, Xie W, Adib E, Stadler WM, Zakharia Y, Alva A, Michaelson MD, Gupta S, Lam ET, Farah S, Nassar AH, Wei XX, Kilbridge KL, Harshman L, Signoretti S, Sholl L, Kwiatkowski DJ, McKay RR, Choueiri TK. Biomarker-Based Phase II Study of Sapanisertib (TAK-228): An mTORC1/2 Inhibitor in Patients With Refractory Metastatic Renal Cell Carcinoma. JCO Precis Oncol. 2022 Feb;6:e2100448. doi: 10.1200/PO.21.00448. PMID 35171658

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 39 patients were enrolled from 8 institutions between August 2017 and November 2019.
Pre-assignment Details: 1 patient was deemed as ineligible and did not receive protocol treatment. 38 eligible and treated patients were included in the analysis.
Groups:
- TAK-228: Subjects will receive treatment with TAK-228 30mg by mouth weekly on day 1, 8, 15 and 22 of a 28-day cycle. Dose can be reduced by the study team. Treatment will continue until disease progression, unaccepted toxicity or other reasons for discontinuation defined by protocol.
Period: Overall Study
Arm/Group | TAK-228
Started | 39
Treated | 38
Completed | 0
Not Completed | 39
Not completed — Still on Therapy | 2
Not completed — Progressive Disease | 29
Not completed — Adverse Event | 4
Not completed — Withdrawal by Subject | 1
Not completed — Physician Decision | 1
Not completed — Patient Decision | 1
Not completed — Ineligible for Study Drug | 1

BASELINE CHARACTERISTICS:
Population: Baseline data was assessed in 38 eligible and treated patients. 1 patient who was deemed as ineligible and did not receive treatment was excluded from baseline analysis.
Groups:
- TAK228: Subjects will receive treatment with TAK-228 30mg by mouth weekly on day 1, 8, 15 and 22 of a 28-day cycle. Dose can be reduced by the study team. Treatment will continue until disease progression, unaccepted toxicity or other reasons for discontinuation defined by protocol.
Arm/Group | TAK228
Number analyzed (Participants) | 38
Age, Continuous [Median (Full Range); unit: years] | 62 [28 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 33
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 36
  More than one race | 2
  Unknown or Not Reported | 0
Histology [Count of Participants; unit: Participants]
  Clear cell histology | 28
  Non clear cell histology | 10
Prior rapalogs treatment [Count of Participants; unit: Participants]
  No | 21
  Yes | 17

OUTCOME MEASURES:

1. Primary Outcome: Best Overall Response Rate
Description: The best overall response rate is the percentage of participants achieving complete response (CR) or partial response (PR) as the best response recorded on treatment based on Response Evaluation Criteria In Solid Tumors Criteria (RECIST 1.1).
  CR and PR must meet the following lesion criteria without having any new lesions as well:
  Target Lesion:
  (CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm.
  (PR): At least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters.
  Non-Target Lesion:
  (CR): Disappearance of all non-target lesions and normalization of tumor marker level. All lymph nodes must be non-pathological in size (<10 mm short axis).
  Non-CR/Non-Progressive Disease: Persistence of one or more non-target lesion(s) and/or maintenance of tumor marker level above the normal limits. Must have PR in target lesion.
Time Frame: Imaging assessments occurred every eight weeks (2 cycles) for response evaluation. The median number of cycles administered was 2 (range <1-15), thus participants were assessed up to ~14 months.
Population: Best overall response was assessed in 38 eligible and treated patients. 1 patient who was deemed as ineligible and did not receive treatment was excluded from response analysis.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | TAK-228
Number analyzed (Participants) | 38
percentage of participants | 5 [1 to 16]

2. Secondary Outcome: Median Progression Free Survival
Description: Progression free survival (PFS) was defined as time from treatment initiation to radiographic progression, clinical progression or death from any cause, or it was censored at the date of last disease evaluation if an event had not occurred. Median PFS was estimated from the Kaplan Meier methodology.
  Radiographic progression is defined by Response Evaluation Criteria In Solid Tumors Criteria 1.1 as follows:
  - >20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (including baseline if it's the smallest).
  OR
  -Appearance of one or more new lesions and/or unequivocal progression of existing non-target lesions.
Time Frame: Participants followed for up to 14 months
Population: Progression free survival was assessed in 38 eligible and treated patients. 1 patient who was deemed as ineligible and did not receive treatment was excluded from analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | TAK-228
Number analyzed (Participants) | 38
months | 2.5 [1.8 to 3.7]

3. Secondary Outcome: Median Overall Survival
Description: Overall survival was defined as the time from treatment initiation to death from any cause or censored at the time of last follow-up for surviving patients. Median overall survival was estimated using the Kaplan Meier methodology.
Time Frame: Participants were follow for up to ~27 months
Population: Overall survival was assessed in 38 eligible and treated patients. 1 patient who was deemed as ineligible and did not receive treatment was excluded from analysis.
Measure: Median (Full Range); unit: months
Arm/Group | TAK-228
Number analyzed (Participants) | 38
months | 11.2 [1 to 27.4]

4. Secondary Outcome: Percentage of Participants With Any Grade 3 or Higher Treatment-related Adverse Events
Description: Toxicity was assessed by Common Terminology Criteria for Adverse Events (CTCAE) version 4.0. Treatment related adverse events were those that were deemed as "Definitely", "Probably" and "Possibly" related to the study treatment.
Time Frame: Adverse events are measured continuously on treatment and up to thirty days after going off treatment (up to ~15 months).
Population: Adverse events were assessed in 38 eligible and treated patients. 1 patient who was deemed as ineligible and did not receive treatment was excluded from analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | TAK-228
Number analyzed (Participants) | 38
Participants
  Number of subjects who experienced grade 3 or higher adverse events | 12
  Number of subjects who did not experience grade 3 or higher adverse events | 26

ADVERSE EVENTS:
Time Frame: Adverse events were assessed from registration to 30 days after end of treatment, up to 15 months. All-Cause Mortality assessed up to approximately 27 months
Description: Serious AEs (SAE) were defined as events with treatment-attribution of possibly, probably or definitely and grade 3 or higher. Remaining AEs are classified as Other AEs (OAE). Maximum grade toxicity by type was calculated within SAE and OAE datasets.
Arm/Group | TAK-228
All-Cause Mortality (participants affected / at risk) | 15/38
Serious Adverse Events (participants affected / at risk) | 12/38
Other Adverse Events (participants affected / at risk) | 38/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TAK-228 (N=38)
Myocardial infarction (Cardiac disorders) | 1
Mucositis oral (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 2
Anorexia (Metabolism and nutrition disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 2
Hyperglycemia (Metabolism and nutrition disorders) | 2
Hyperkalemia (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1
Chronic kidney disease (Renal and urinary disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1
Vascular disorders - Other, specify (Vascular disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TAK-228 (N=38)
Anemia (Blood and lymphatic system disorders) | 9
Leukocytosis (Blood and lymphatic system disorders) | 1
Lymph node pain (Blood and lymphatic system disorders) | 1
Atrioventricular block first degree (Cardiac disorders) | 1
Chest pain - cardiac (Cardiac disorders) | 1
Palpitations (Cardiac disorders) | 1
Sinus bradycardia (Cardiac disorders) | 1
Sinus tachycardia (Cardiac disorders) | 2
Cardiac disorders - Other, specify (Cardiac disorders) | 2
Tinnitus (Ear and labyrinth disorders) | 1
Adrenal insufficiency (Endocrine disorders) | 1
Hyperparathyroidism (Endocrine disorders) | 1
Hyperthyroidism (Endocrine disorders) | 1
Hypothyroidism (Endocrine disorders) | 4
Endocrine disorders - Other, specify (Endocrine disorders) | 1
Eye pain (Eye disorders) | 1
Retinal detachment (Eye disorders) | 1
Watering eyes (Eye disorders) | 1
Abdominal distension (Gastrointestinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 3
Anal pain (Gastrointestinal disorders) | 1
Colitis (Gastrointestinal disorders) | 2
Constipation (Gastrointestinal disorders) | 15
Diarrhea (Gastrointestinal disorders) | 9
Dry mouth (Gastrointestinal disorders) | 4
Duodenal hemorrhage (Gastrointestinal disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 2
Gastroesophageal reflux disease (Gastrointestinal disorders) | 4
Mucositis oral (Gastrointestinal disorders) | 12
Nausea (Gastrointestinal disorders) | 26
Small intestinal obstruction (Gastrointestinal disorders) | 1
Stomach pain (Gastrointestinal disorders) | 1
Toothache (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 13
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 3
Chills (General disorders) | 3
Edema limbs (General disorders) | 4
Fatigue (General disorders) | 24
Fever (General disorders) | 2
Gait disturbance (General disorders) | 1
Non-cardiac chest pain (General disorders) | 3
Pain (General disorders) | 7
General disorders and administration site conditions - Other, specify (General disorders) | 3
Bile duct stenosis (Hepatobiliary disorders) | 1
Nail infection (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 1
Upper respiratory infection (Infections and infestations) | 2
Urinary tract infection (Infections and infestations) | 2
Vaginal infection (Infections and infestations) | 1
Bruising (Injury, poisoning and procedural complications) | 1
Fracture (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 2
Aspartate aminotransferase increased (Investigations) | 2
Blood bilirubin increased (Investigations) | 1
Cholesterol high (Investigations) | 2
Creatinine increased (Investigations) | 6
Lymphocyte count decreased (Investigations) | 1
Platelet count decreased (Investigations) | 3
Weight loss (Investigations) | 1
Investigations - Other, specify (Investigations) | 1
Anorexia (Metabolism and nutrition disorders) | 16
Dehydration (Metabolism and nutrition disorders) | 4
Hypercalcemia (Metabolism and nutrition disorders) | 2
Hyperglycemia (Metabolism and nutrition disorders) | 5
Hyperkalemia (Metabolism and nutrition disorders) | 7
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 2
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 1
Abdominal soft tissue necrosis (Musculoskeletal and connective tissue disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 8
Bone pain (Musculoskeletal and connective tissue disorders) | 2
Buttock pain (Musculoskeletal and connective tissue disorders) | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 5
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 2
Amnesia (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 2
Dysgeusia (Nervous system disorders) | 2
Headache (Nervous system disorders) | 4
Memory impairment (Nervous system disorders) | 1
Peripheral motor neuropathy (Nervous system disorders) | 1
Seizure (Nervous system disorders) | 1
Tremor (Nervous system disorders) | 2
Nervous system disorders - Other, specify (Nervous system disorders) | 1
Agitation (Psychiatric disorders) | 1
Anxiety (Psychiatric disorders) | 1
Confusion (Psychiatric disorders) | 1
Delirium (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 2
Insomnia (Psychiatric disorders) | 3
Suicidal ideation (Psychiatric disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 3
Hematuria (Renal and urinary disorders) | 2
Hemoglobinuria (Renal and urinary disorders) | 1
Proteinuria (Renal and urinary disorders) | 2
Urinary frequency (Renal and urinary disorders) | 3
Urinary retention (Renal and urinary disorders) | 1
Urinary tract obstruction (Renal and urinary disorders) | 1
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 4
Breast pain (Reproductive system and breast disorders) | 1
Apnea (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 10
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 7
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 4
Tracheal fistula (Respiratory, thoracic and mediastinal disorders) | 1
Bullous dermatitis (Skin and subcutaneous tissue disorders) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 2
Pruritus (Skin and subcutaneous tissue disorders) | 5
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 9
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 3
Surgical and medical procedures - Other, specify (Surgical and medical procedures) | 1
Hematoma (Vascular disorders) | 2
Hypertension (Vascular disorders) | 1
Hypotension (Vascular disorders) | 5
Thromboembolic event (Vascular disorders) | 1
Vascular disorders - Other, specify (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-12-20): https://cdn.clinicaltrials.gov/large-docs/28/NCT03097328/Prot_SAP_000.pdf